CLINICAL TRIAL: NCT06013124
Title: Organizational Environment, Staff Well-being and Patient/Caregiver Perceived Quality of Care in a Maternal and Child Health Hospital in Italy
Brief Title: Patient/Caregiver Perceived Quality of Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 46/20
Record Dates: First submitted 2023-03-24; First posted 2023-08-28 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2023-08

CONDITIONS: Maternal and Child Health
Keywords: Patient safety; occupational health; health care quality assurance
MeSH Terms: interventions — Working Conditions; Health

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Work environment, well-being, customer satisfaction — Evaluation hospital work environment, staff well-being features and patients/caregivers satisfaction and perceived quality of care

SUMMARY:
Hospitals quality, safety, and staff workload problems are common in all countries. Findings from the multicountry Nurse forecasting in Europe (RN4CAST) cross sectional study show that patient risk of mortality within a 30 days of hospital stay increases of 7% when a patient is added to the nurse-patient 1:6 proportion in a surgical unit; in Italy, the ratio was found to be 9.5 patients per nurse. Organizational environment, health workers wellbeing and work satisfaction were also found to impact patient safety and perceived patient satisfaction; hospitals nurses high workload, work dissatisfaction and burnout were found related to poor patients outcomes. In a systematic review and meta-analysis, an association of more than 60% between physicians and nurses development of burnout and patient safety in pediatric settings was found; when health workers wellness and teamwork in wards was poor lower perceptions of safety culture was found. Moreover, occupational exposure to medically complex children and their families along with direct care providers unexpressed grief further increase pediatric settings staff risk of developing burnout syndrome and compassion fatigue. Recent findings of Covid-19 pandemic negative impact on health workers well-being worldwide also enhances the risk of compromising the quality of care provided. The aim of this study is to evaluate factors that affect health workers well-being, their perception of work environment and patient/caregiver satisfaction and perceived quality of care in a maternal and child health hospital.

ELIGIBILITY:
Inclusion Criteria:

* Health workers directly involved in patients care and employed for more than 6 months
* Patients (adults, school-aged children)
* Caregivers of children

Exclusion Criteria:

* Health workers employed for less than 6 months

Ages: 6 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Health workers, patients (adults and school-aged children), caregivers of children
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Hospital Work environment | Through study completion, an average of 3 year
  Evaluated by validated questionnaire
Staff well-being | Through study completion, an average of 3 year
  Evaluated by validated questionnaire
Patients/caregivers satisfaction | Through study completion, an average of 3 year
  Evaluated by validated questionnaire
Patients/caregivers perceived quality of care | Through study completion, an average of 3 year
  Evaluated by validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Raffaella Raffaella, MSC, Principal Investigator — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided